CLINICAL TRIAL: NCT05057689
Title: A Double-blinded, Randomized Trial Comparing the Safety & Efficacy of Intranasal Dexmedetomidine, Intranasal Fentanyl & Intranasal Midazolam in the Pediatric Emergency Room
Brief Title: Safety & Efficacy of Intranasal Dexmedetomidine, Fentanyl & Midazolam in the Pediatric Emergency Room
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Unable to obtain funding to initiate/complete study
Sponsor: Nationwide Children's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 261081
Record Dates: First submitted 2021-09-15; First posted 2021-09-27 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Acute Stress Disorder; Anxiety; Pain
MeSH Terms: conditions — Stress Disorders, Traumatic, Acute; Anxiety Disorders; Pain | interventions — Dexmedetomidine; Fentanyl

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Intranasal Dexmedetomidine (4 mcg/kg) (Experimental): Dexmedetomidine 100 mcg/mL (concentration of 200 mcg/2 mL) will be atomized for intranasal administration at a dose of 4 mcg/kg (0.04 mL/kg) according to a weight-based dosing chart. The maximum dose will be 200 mcg.
  Interventions: Drug: Intranasal Dexmedetomidine (4 mcg/kg)
- Intranasal Fentanyl (2 mcg/kg) (Experimental): Fentanyl 50 mcg/mL (concentration of 100 mcg/2 mL) will be atomized for intranasal administration at a dose of 2 mcg/kg (0.04 mL/kg) according to a weight-based dosing chart. The maximum dose will be 100 mcg.
  Interventions: Drug: Intranasal Fentanyl (2 mcg/kg)
- Intranasal Midazolam (5 mg/kg) (Experimental): Midazolam 5 mg/mL (concentration of 10 mg/2 mL) will be atomized for intranasal administration at a dose of 0.3 mg/kg (0.06 mL/kg) according to a weight-based dosing chart. The maximum dose will be 10 mg
  Interventions: Drug: Intranasal Midazolam (5 mg/kg)

INTERVENTIONS:
Drug: Intranasal Dexmedetomidine (4 mcg/kg) — Dexmedetomidine 100 mcg/mL (concentration of 200 mcg/2 mL) will be atomized for intranasal administration at a dose of 4 mcg/kg (0.04 mL/kg) according to a weight-based dosing chart prior to laceration repair. The maximum dose will be 200 mcg.
  Other Names: Precedex
  Arms: Intranasal Dexmedetomidine (4 mcg/kg)
Drug: Intranasal Fentanyl (2 mcg/kg) — Fentanyl 50 mcg/mL (concentration of 100 mcg/2 mL) will be atomized for intranasal administration at a dose of 2 mcg/kg (0.04 mL/kg) according to a weight-based dosing chart prior to laceration repair. The maximum dose will be 100 mcg.
  Other Names: Fentanyl Citrate
  Arms: Intranasal Fentanyl (2 mcg/kg)
Drug: Intranasal Midazolam (5 mg/kg) — Midazolam 5 mg/mL (concentration of 10 mg/2 mL) will be atomized for intranasal administration at a dose of 0.3 mg/kg (0.06 mL/kg) according to a weight-based dosing chart prior to laceration repair. The maximum dose will be 10 mg.
  Arms: Intranasal Midazolam (5 mg/kg)

SUMMARY:
The hypothesis is that intranasal dexmedetomidine will provide significantly more effective analgesia and anxiolysis for subjects undergoing a simple laceration repair when compared to either intranasal fentanyl or intranasal midazolam.

Additional hypotheses include that there will be 1) no significant increase in adverse effects between drugs and 2) significantly higher satisfaction rates for both subject experience and ease of laceration repair based on structured, proceduralist feedback.

DETAILED DESCRIPTION:
Intranasal medications are rapidly gaining popularity as agents for analgesia and anxiolysis in the pediatric hospital setting. One of the primary reasons for the popularity of intranasal medications is ease of administration combined with favorable pharmacokinetics. It has been well established that children identify venipuncture as one of the most painful and anxiety-producing procedures during time spent in the hospital, and these experiences have been shown to have a more lasting impact, producing increased anxiety and fear at subsequent visits. Although oral and rectal administration of analgesics are also non-invasive, bioavailability, time to onset, and half-lives are significantly longer with these routes of administration in comparison to intranasal administration. Multiple studies have shown that intranasal fentanyl, midazolam, and dexmedetomidine have similar pharmacokinetics to intravenous preparations and reach adequate serum levels in both the blood and cerebrospinal fluid. In the pediatric emergency room setting, intranasal fentanyl and midazolam have been shown to provide effective analgesia and anxiolysis for a variety of settings, including pain management (e.g. pain associated with long bone fractures, burns, incision and drainage) and pre-procedural sedation/anxiolysis (e.g. radiological imaging).Numerous studies have examined the safety and efficacy of intranasal fentanyl and midazolam, and several studies have examined the efficacy of intranasal dexmedetomidine for non-painful procedural sedation. To date, two studies have compared the use of intranasal dexmedetomidine and intranasal midazolam or intranasal dexmedetomidine, intranasal fentanyl, and intranasal midazolam for anxiolysis in painful procedural sedations. However, as of 2020, no previous studies have compared the use of intranasal dexmedetomidine, intranasal fentanyl, and intranasal midazolam for painful procedures in the pediatric emergency setting.

ELIGIBILITY:
Inclusion Criteria:

* Primary complaint of "laceration"
* 2 years to 6 years of age (inclusive)
* Initial presentation at the Arkansas Children's Hospital (ACH) Emergency Department

Exclusion Criteria:

* Prior allergic reaction to fentanyl or midazolam or dexmedetomidine
* Prior major adverse reaction to fentanyl or midazolam (e.g. seizure-like activity, paradoxical reaction, hallucinations)
* Nasal injury/deformity
* Potential for altered pain perception (e.g. autism, severe sensory-neural disturbances)
* History of adverse reaction to sedation/anesthesia
* History of cardiac arrhythmia
* History of liver dysfunction
* Concurrent injuries that would necessitate higher levels of care (e.g. inpatient admission, immediate evaluation in the operating room (OR), etc.)
* Complex (multi-layer) lacerations or those requiring subspecialty consultation for repair
* American Society of Anesthesiology (ASA) score ≥ 3
* Use of analgesics (with the exception of ibuprofen or acetaminophen) or anxiolytics in the immediate pre-examination period (within 4 hours)

Ages: 2 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2025-09 (Estimated); Primary Completion 2025-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Pain using the Face, Legs, Activity, Cry, Consolability (FLACC) scale | through the procedure, an average of 1 day
  Analgesia in subjects undergoing simple laceration repair will be compared across the three investigational drug products (intranasal dexmedetomidine, intranasal fentanyl, and intranasal midazolam) using the FLACC scale.
Anxiety using the modified Yale Preoperative Anxiety Scale (mYPAS) behavior observation tool | through the procedure, an average of 1 day
  Anxiolysis in subjects undergoing simple laceration repair will be compared across the three investigational drug products (intranasal dexmedetomidine, intranasal fentanyl, and intranasal midazolam) using the modified Yale Preoperative Anxiety Scale (mYPAS) behavior observation tool.

SECONDARY OUTCOMES:
Satisfaction rates for subject experience across the three study drugs based on parent/legally authorized representative (LAR) survey | within 1 week of the laceration repair, average of 5 days
  Parent/LAR will be asked to complete a follow-up survey so that parent/LAR can provide feedback on the level of satisfaction with the laceration repair experience.
Satisfaction rates for surgical repair across the three study drugs based on proceduralist survey | within 1 week of the laceration repair, average of 5 days
  Proceduralist will be asked to complete a follow-up survey to provide feedback on the level of satisfaction with the laceration repair experience.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Chang, MD, Principal Investigator — University of Arkansas
Locations (1):
- Arkansas Children's Hospital, Little Rock, Arkansas, United States